CLINICAL TRIAL: NCT00196508
Title: A Randomized, Multi Center Study to Evaluate the Clinical Performance of Topical Skin Adhesive in Comparison to Sutures for Perineal Skin Closure Following Childbirth
Brief Title: A Study Comparing Topical Skin Adhesive or Sutures for Closure Due to Episiotomy or Perineal Tears Following Childbirth
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 200-04-001
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2007-10-16 (Estimated); Status verified 2006-06

CONDITIONS: Episiotomy; Perineal Tear
Keywords: Childbirth

INTERVENTIONS:
Device: High Viscosity DERMABOND

SUMMARY:
This is a randomized controlled trial and multi-centered study with a 2-arm design. The treatment group will receive topical skin adhesive for skin closure of their wound and the control will receive sutures. Subjects will be assessed at follow-up visits. Patients are required to maintain a diary postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age.
* Patient has an episiotomy incision or perineal tear resulting from a vaginal delivery.
* Patient agrees to participate in the follow-up schedule of assessments and completion of a daily diary.
* Patient has signed the informed consent form.

Exclusion Criteria:

* Patient has peripheral vascular disease.
* Patient has insulin dependent diabetes mellitus.
* Patient has a blood clotting disorder that requires therapy.
* Patient has a personal or family history of keloid formation or hypertrophy.
* Patient has a known allergy to cyanoacrylates or formaldehyde.
* Patient has impaired wound healing by history. Patient is a chronic steroid user.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118
Dates: Start 2005-04; Study Completion 2006-01

PRIMARY OUTCOMES:
Topical skin adhesive is non-inferior to sutures when used for skin closure following an episiotomy incision or perineal tear resulting from childbirth
The incidence of perineal skin opening requiring re-closure post-partum

SECONDARY OUTCOMES:
Presence and extent of clinically relevant skin openings
Presence and extent of acute inflammatory reaction, pain, itch and discomfort associated with the perineal skin area
Perineal skin closure cosmesis
Patient satisfaction

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Bessemer, Alabama
  - Phoenix OB-GYN Associates, Moorestown, New Jersey
  - McDonald Murrmann Women's Clinic, Memphis, Tennessee
  - Tidewater Physicians for Women, Norfolk, Virginia
  - Virginia Beach Obstetrics & Gynecology, Virginia Beach, Virginia